CLINICAL TRIAL: NCT01348724
Title: A Phase I, Open-Label, Single-Centre Study to Assess Absorption, Distribution, Metabolism and Excretion (ADME) After [14C]-Labelled Oral Administration of NKTR-118 to Healthy Male Volunteers
Brief Title: Absorption, Distribution, Metabolism and Excretion (ADME) Study With Single Oral Administration of [14C] NKTR-118
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D3820C00001
Record Dates: First submitted 2011-04-21; First posted 2011-05-05 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Volunteers
Keywords: Radioactive carbon; Absorption; Distribution; Metabolism; Excretion; Healthy Volunteers
MeSH Terms: interventions — naloxegol

ARMS (1):
- [14C] NKTR-118 (Experimental)
  Interventions: Drug: [14C] NKTR-118

INTERVENTIONS:
Drug: [14C] NKTR-118 — Single 25 mg oral dose administered on Day 1

SUMMARY:
Study to Assess the Absorption, Metabolism and Excretion of [14C] NKTR-118 after a Single-Dose Oral Administration.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of ≥18 and ≤30 kg/m2 and a minimum weight of 50 kg
* Regular daily bowel movements (ie, production of at least 1 stool per day).
* Non-smoker or ex-smoker who has not used tobacco or nicotine products for ≥3 months prior to Visit 1

Exclusion Criteria:

* Healthy volunteers who have been exposed to radiation levels above background (eg, through X-ray examination) of >5 mSv in the last year, >10 mSv in the last 5 years, or a cumulative total of >1 mSv per year of life
* Participation in any prior radiolabelled study within 12 months of screening visit 1
* Excessive intake of caffeine containing drinks e.g., coffee, tea, caffeine containing energy drinks and cola (more than 5 cups of coffee or equivalent per day

Ages: 35 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Percentage of radioactive dose recovered in urine and feces samples and the total percentage of radioactive dose recovered in both urine and feces | Range of Day 1 until day 10
Concentration of total radioactivity in blood and plasma samples | Range of Day 1 until day 10
Concentration of NKTR-118 in blood and plasma sample | Range of Day 1 until day 10

SECONDARY OUTCOMES:
Safety and tolerability of NKTR-118 following administration of a single oral dose of [14] NKTR-118 solution by assessing adverse event | Range of Day -1 until follow up visit (Visit 3)
Safety and tolerability of NKTR-118 following administration of a single oral dose of [14] NKTR-118 solution by assessing vital signs | Range of Day -1 until follow up visit (Visit 3)
Safety and tolerability of NKTR-118 following administration of a single oral dose of [14] NKTR-118 solution by assessing safety blood samples | Range of Day -1 until follow up visit (Visit 3)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Kasti, MD, Principal Investigator — Quintiles, Inc.; Mark Sostek, PhD, Study Director — AstraZeneca; Emeline Ramos, Study Chair — AstraZeneca
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- See also: Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1385&filename=D3820C00001_Clinical_Study_Report_Synopsis.pdf